CLINICAL TRIAL: NCT01236807
Title: MR INFORM - a Randomized Non-inferiority Multicenter Trial Comparing MR Perfusion Imaging and Fractional Flow Reserve (FFR) to Guide Management of Patients With Stable Coronary Artery Disease
Brief Title: MR INFORM - MR Perfusion Imaging to Guide Management of Patients With Stable Coronary Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other); Bayer (Industry)
Responsible Party: Principal Investigator, Eike Nagel, Global Chief Investigator, King's College London
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: MR INFORM-10
Record Dates: First submitted 2010-11-08; First posted 2010-11-09 (Estimated); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Coronary Artery Disease; Stable Angina; Myocardial Ischaemia
Keywords: Adenosine; Magnetic Resonance Imaging; MR perfusion; Fractional Flow Reserve, Myocardial; FFR; Pressure wire; Coronary Disease; Heart Diseases; Cardiovascular Diseases; Arteriosclerosis
MeSH Terms: conditions — Coronary Artery Disease; Angina, Stable; Coronary Disease; Heart Diseases; Cardiovascular Diseases; Arteriosclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MR Inform (Active Comparator): Management guided by the result of the MR perfusion scan. Possible intervention: coronary artery revascularization.
  Interventions: Procedure: MR perfusion guidance
- FFR Inform (Active Comparator): Management guided by the result of FFR measurement. Possible intervention: coronary artery revascularization.
  Interventions: Procedure: FFR guidance

INTERVENTIONS:
Procedure: MR perfusion guidance — Coronary revascularization guided by MR perfusion imaging
  Arms: MR Inform
Procedure: FFR guidance — Coronary revascularization guided by invasive angiography and FFR
  Arms: FFR Inform

SUMMARY:
The purpose of this study is to determine if MR Perfusion Imaging is non-inferior to coronary angiography with measurement of Fractional Flow Reserve (FFR) in guiding management of patients with stable chest pain.

* All patients will undergo an MR Perfusion Imaging test.
* Further management will be guided by the result of the cardiac MRI in half of the patients (chosen by random).
* The other half will undergo coronary angiography with measurement of FFR. The result of this test alone will guide their further management. The result of the initial MR Perfusion test will not be available to the treating doctors of this group.
* All patients will receive optimal medical therapy (OMT)
* All patients will undergo follow-up to find out if they have any relevant heart related events.

ELIGIBILITY:
Inclusion Criteria:

* Angina pectoris CCS class II and III and either
* ≥2 cardiovascular risk factors
* or positive exercise treadmill test
* Signed written informed consent
* age: at least 18 years

Exclusion Criteria:

* contraindication to MR
* contraindication to adenosine infusion
* EF≤ 30%
* inability to lie supine for 60 minutes
* previous Coronary Artery Bypass Grafts
* revascularization within the previous 6 months
* cardiac arrhythmias (atrial fibrillation, >20 ectopic beats/min)
* poor renal function (eGFR <30ml/min)
* body weight > 140kg or waist perimeter > 95cm
* known allergy to contrast media

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 915 (Actual)
Dates: Start 2010-12; Primary Completion 2016-08 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Occurence of major adverse cardiac events (MACE) | 1year
  Composite of all cause death, myocardial infarction and repeat revascularisation.

SECONDARY OUTCOMES:
Individual MACE | 1 year
  individual components as defined above
Other adverse events | 1 year
  need for revascularization after initial treatment within 1 year
Course of symptoms (angina, breathlessness) | 1 year
  CCS class, NYHA class
Cost comparison | 1 year
  Costs related to MR- and FFR-guided selection for revascularisation
changes in LV volumes and function | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Eike Nagel, MD, PhD, Principal Investigator — Goethe University Frankfurt
Locations (1):
- King's College, London, United Kingdom

REFERENCES:
- [Background] Hussain ST, Paul M, Plein S, McCann GP, Shah AM, Marber MS, Chiribiri A, Morton G, Redwood S, MacCarthy P, Schuster A, Ishida M, Westwood MA, Perera D, Nagel E. Design and rationale of the MR-INFORM study: stress perfusion cardiovascular magnetic resonance imaging to guide the management of patients with stable coronary artery disease. J Cardiovasc Magn Reson. 2012 Sep 19;14(1):65. doi: 10.1186/1532-429X-14-65. PMID 22992411
- [Background] Nagel E, Berry C. Magnetic Resonance Perfusion or Fractional Flow Reserve in Coronary Disease. Reply. N Engl J Med. 2019 Dec 5;381(23):2277-2278. doi: 10.1056/NEJMc1913968. No abstract available. PMID 31801003
- [Result] Nagel E, Greenwood JP, McCann GP, Bettencourt N, Shah AM, Hussain ST, Perera D, Plein S, Bucciarelli-Ducci C, Paul M, Westwood MA, Marber M, Richter WS, Puntmann VO, Schwenke C, Schulz-Menger J, Das R, Wong J, Hausenloy DJ, Steen H, Berry C; MR-INFORM Investigators. Magnetic Resonance Perfusion or Fractional Flow Reserve in Coronary Disease. N Engl J Med. 2019 Jun 20;380(25):2418-2428. doi: 10.1056/NEJMoa1716734. PMID 31216398